CLINICAL TRIAL: NCT05675228
Title: Knowledge of Young Adults About Genital Herpes
Acronym: HerpesG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_RIPH_016_HerpesG
Record Dates: First submitted 2022-12-29; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Genital Herpes
Keywords: Knowledge; Young adults; genital herpes
MeSH Terms: conditions — Herpes Genitalis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- young adults: men and women aged 25 to 35
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Knowledge about genital herpes

SUMMARY:
Despite sex education in schools and prevention campaigns concerning sexually transmitted infections, genital herpes remains frequent infection. In 2016, according to the World Health Organization, more than 490 million people worldwide were living with a genital herpes infection.

DETAILED DESCRIPTION:
the aim of the study is to describe knowledge of adults aged 25 to 35 about genital herpes (symptoms, transmission, prevention).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 25 to 35
* Having sex or not
* Agreeing to participate in the study

Exclusion Criteria:

- Not agreeing to participate in this study

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: men and women aged 25 to 35, having sex or not and agreeing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
transmission | Day 0
  Modes of transmission of genital herpes (public toilets, home textiles, sexual transmission)
symptoms | Day 0
  Types of symptoms of genital herpes (no symptom, rash, fever)

CONTACTS AND LOCATIONS:
Locations (1):
- Fanny Bichon, Reims, France